CLINICAL TRIAL: NCT04957160
Title: A Multicentre, Retrospective, Non-interventional Review of Electronic Prescribing Records of Any Second-line (2L) Patients and Chart Notes of 2L Cabozantinib Patients, Investigating the Treatment Sequence Pathway Following a First-line, Immuno-oncology Checkpoint Inhibitor (1L IO) Containing Combination Therapy in Patients With Advanced Renal Cell Carcinoma (aRCC) (CARINA)
Brief Title: Cabozantinib Post First-line Immuno-oncology Checkpoint Inhibitor Containing Combination
Acronym: CARINA
Status: Completed | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60000-451
Record Dates: First submitted 2021-01-12; First posted 2021-07-12 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Advanced Renal Cell Carcinoma (aRCC)

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1
- Cohort 2

SUMMARY:
This study will collect real-world data for the new treatment pathways for all patients with Advanced Renal Cell Carcinoma (ARCC) who were treated with a 1L IO (first-line, Immuno-Oncology checkpoint inhibitor) combination therapy and progressed to a 2L treatment with particular focus to understanding where cabozantinib is prescribed after 1L IO containing combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of aRCC.
* Patients aged ≥18 years at aRCC diagnosis treated with a 1L IO containing combination therapy who have progressed to a 2L treatment.

Exclusion Criteria:

* Patient's hospital medical records are unavailable for review;
* Patients have started a 2L treatment as part of a Renal Carcinoma Treatment (RCT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in 10 UK hospitals that have patients who have been treated with a 1L IO containing combination therapy and have progressed to, and started, a 2L treatment.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Description of the treatment sequence pathway from 1L up to 2L for patients with aRCC | From start of treatment to last hospital follow-up or date of death whichever occurs first assessed during data collection period (from 15th of January 2015 until September 2022)
  To be described for patients with aRCC receiving 2L treatment following a 1L IO containing combination therapy.
Description of the treatment sequence pathway from 1L up to the 2L for cabozantinib patients with aRCC | From start of treatment to last hospital follow-up or date of death whichever occurs first assessed during data collection period (from 15th of January 2015 until September 2022)
  To be described for patients with aRCC receiving 2L treatment and subsequent lines of treatment following a 1L IO containing combination therapy.

SECONDARY OUTCOMES:
Overall Survival (OS) | From start of treatment to last hospital follow-up or date of death whichever occurs first assessed during data collection period (from 15th of January 2015 until September 2022)
Time to Treatment Discontinuation (TTD) by line | From start date of first cycle of treatment to start date of last cycle of treatment during data collection period (from 15th of January 2015 until September 2022)
Physician defined Best Response by line - complete response, partial response, stable disease, progressive disease | From start of treatment to last hospital follow-up or date of death whichever occurs first assessed during data collection period (from 15th of January 2015 until September 2022)
Overall Response Rate (ORR) by line -complete response or partial response | From start of treatment to last hospital follow-up or date of death whichever occurs first assessed during data collection period (from 15th of January 2015 until September 2022)
Duration of treatment by line | From start date of first cycle of treatment to start date of last cycle of treatment during data collection period (from 15th of January 2015 until September 2022)
Drug start and end dose by line | From start of treatment to last hospital follow-up or date of death whichever occurs first assessed during data collection period (from 15th of January 2015 until September 2022)
  Descriptive statistics using following parameters: no dose change, dose change, dose increase and dose decrease
Disease Control Rate (DCR) by line - complete response, partial response and stable disease | From start of treatment to last hospital follow-up or date of death whichever occurs first assessed during data collection period (from 15th of January 2015 until September 2022)
Progression Free Survival (PFS) by line for cabozantinib patients | From start of treatment to last hospital follow-up or date of death whichever occurs first assessed during data collection period (from 15th of January 2015 until September 2022)
Reason for stopping cabozantinib | From start of treatment to last hospital follow-up or date of death whichever occurs first assessed during data collection period (from 15th of January 2015 until September 2022)
  Descriptive statistics using the following parameters: radiological disease progression, clinical deterioration, AE, subject's decision, Investigator's decision, end of predefined treatment, other
Reason for dose change (Disease progression, AE, subject non-compliance, subject decision, clinical / Investigator decision, radiotherapy(s), surgery(s), COVID-19 pandemic, other) | From start of treatment to last hospital follow-up or date of death whichever occurs first assessed during data collection period (from 15th of January 2015 until September 2022)
Describe interruptions for cabozantinib | From start of treatment to last hospital follow-up or date of death whichever occurs first assessed during data collection period (from 15th of January 2015 until September 2022)
Cause of death (RCC or non RCC related) | From start of treatment to last hospital follow-up or date of death whichever occurs first assessed during data collection period (from 15th of January 2015 until September 2022)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (9):
- United Kingdom (9):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Surrey County Hospital, Guildford
  - Barts Cancer Institute, London
  - Royal Marsden Hospital, London
  - Christie NHS Foundation Trust, Manchester
  - Clatterbridge Road, Bebington, Metropolitan Borough of Wirral
  - Nottingham University Hospital, Nottingham
  - Royal Preston Hospital, Preston
  - Mount Vernon Cencer Centre, Welwyn Garden City